CLINICAL TRIAL: NCT02901938
Title: Feasibility of Implantation of Cemented Femoral Stem in the Treatment of Osteoporotic Femoral Neck Fracture in Elderly Patients: a Randomized Controlled Trial
Brief Title: Feasibility of Implantation of Cemented Femoral Stem for Osteoporotic Femoral Neck Fracture in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qinghai University (Other)
Responsible Party: Principal Investigator, Rong, Attending Physician, Qinghai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QinghaiUH_004
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Femoral Neck Fracture
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cemented femoral stem group (Experimental): The patients with avascular necrosis of the femoral head complicated by osteoporotic femoral neck fracture will be randomly assigned to undergo implantation of cemented femoral stem.
  Interventions: Procedure: cemented femoral stem
- cannulated compression screws group (Experimental): The patients with avascular necrosis of the femoral head complicated by osteoporotic femoral neck fracture will be randomly assigned to undergo percutaneous internal fixation with cannulated compression screws.
  Interventions: Device: cannulated compression screws

INTERVENTIONS:
Procedure: cemented femoral stem — The patients assigned even numbers will undergo implantation of cemented femoral stem.
  Arms: cemented femoral stem group
Device: cannulated compression screws — The patients assigned even numbers will undergo percutaneous internal fixation with cannulated compression screws.
  Arms: cannulated compression screws group

SUMMARY:
This study will investigate the effects of implantation of cemented femoral stem versus percutanous internal fixation with cannulated compression screws on hip joint function recovery, pains, femoral head collapse and sterile prosthesis loosening, peri-prosthesis infection, and the histocompatibility of prosthesis material with host tissue in the elderly patients with osteoporotic fracture of proximal femoral neck complicated by avascular necrosis of the femoral head, which will provide scientific evidence for selecting surgical methods and internal fixation/artificial prosthesis material for osteoporotic fracture of proximal femoral neck in the elderly patients.

DETAILED DESCRIPTION:
History and current related studies Femoral neck fracture is a common fracture that accounts for 3.58% of all fractures, easily occurs in the elderly with a gradually increased incidence, predisposes to bone nonunion, and greatly influences patient's mental and physical health. Bone nonunion easily occurs after femoral neck fracture because of anatomic position, biomechanical property and local blood supply. The objective of treatment of femoral neck fracture in patients aged 65 years and above is to rapidly restore lower limb function and reduce the complications caused by long term bed rest. Surgery for treatment of femoral neck fracture in the elderly is a satisfactory option because it not only contributes to recovery of joint function, but also decreases the incidence of complications. Several concerns are addressed during the process from design of internal fixation equipment to selection of clinical treatment protocol including minimizing surgical trauma, shortening length of surgery, and promoting functional recovery of hip joint. Osteoporosis is generally considered the most difficult problem to be solved after surgery for femoral neck fracture in the elderly patients. The key points of internal fixation for femoral neck fracture are to optimize bone space and strengthen fractured bone trabecula, yielding strong fixation biomechanically. Percutaneous internal fixation with cannulated compression screws has become a preferred treatment method of osteoporotic femoral neck fracture in elderly patients because of its short length of surgery and less blood loss, but insufficient holding power of used screws in the femoral neck cannot lead to strong fixation. Therefore, joint prosthesis is recommended for repair of femoral neck fracture in elderly patients. Implantation of femoral stem for treatment of early proximal femoral neck fracture has achieved confirmed clinical efficacy, but the long-term therapeutic effects in the treatment of osteoporotic fracture of proximal femoral neck remain poorly understood in patients with avascular necrosis of the femoral head.

Novelty of this study The investigators performed a search of PubMed, Web of Science and Wanfang Database up to August 2016 for articles regarding artificial prosthesis treatment of osteoporotic femoral neck fracture and found that the majority of previous reports focused on early femoral neck fracture and patients were generally followed up no more than 6 months. In this study, we will for the first time investigate the feasibility of implantation of cemented femoral stem versus percutaneous internal fixation with cannulated compression screws in the treatment of osteoporotic femoral neck fracture in the elderly patients with avascular necrosis of the femoral head necrosis through a 12 month follow up observation in terms of hip joint function, pain, histocompatibility of biomaterial with host tissue, and postoperative complications.

Data collection, management, analysis and open access An electronic data capture (EDC) system will be used for data collection and management. All study data will be in time recorded on the electronic case report form provided by the sponsor after patient's visits for recheck unless the outcomes cannot be achieved immediately. Thus, the recorded information can reflect patient's latest outcomes. Information accuracy will be rechecked after all included patients are followed up. The electronic data capture system will be locked by the project manager and will not be altered. All information relating to this trial will be preserved by Qinghai University Affiliated Hospital. The electronic data will be fully disclosed to a professional statistician for statistical analysis. Anonymized trial data will be published at http: www.figshare.com.

Statistical analysis Normally distributed continuous variables will be expressed as the mean ±SD and non-normally distributed variables will be expressed as median and quartile. Categorical variables will be expressed as counts and percentages. All data will be statistically analyzed using SPSS 19.0 software (IBM Corp., Armonk, NU, USA). Two-samples t-test or Mann-Whitney U test will be used for comparisons of Harris hip scores and VAS scores between percutaneous internal fixation with cannulated compression screws and implantation of femoral stem. The chi-square test or Fisher's exact test will be used for comparison of histocompatibility of biomaterial with host tissue. A level of P < 0.05 will be considered statistically significant.

Confidentiality Only the necessary data limited to studying the effectiveness and safety of percutaneous internal fixation with cannulated compression screws/implantation of femoral stem in the treatment of osteoporotic femoral neck fracture in the elderly patients will be collected and processed.

The privacy of information regarding the patients will be safeguarded during data collection and processing, and related laws and regulations should be abided by as follows:

* The process of data collection is fair and legal.
* The objective of data collection is specialized, identified and legal.
* The collected data are abundant, relative but not excessive to the study objective, and the data unrelated to study objective will not be collected.
* The collected data are accurate and will be updated if necessary.
* Consent regarding data collection will be acquired before data collection.
* The collected data will not be disclosed to any non-authorized persons or unlawfully mistaken, lost or altered. During the whole study period, the sponsor persons who have the rights to read the patient's information will not disclose the information.

Advantages and limitations of this study Advantages: This is a prospective, randomized controlled, open-label trial, in which we will evaluate the feasibility of percutaneous internal fixation with cannulated compression screws and implantation of cemented femoral stem in the treatment of osteoporotic femoral neck fracture complicated by avascular necrosis of the femoral head in the elderly patients through evaluating the safety and efficacy of these two surgical methods. In addition, scant information is reported on the biocompatibility of implants with host tissue in patients with osteoporotic femoral neck fracture in the elderly patients. Therefore, our findings will fill the gap.

Limitations: Quality of life and daily activities are also important indices used to evaluate the efficacy of surgery. But this study will be limited to human and material sources, so evaluations on but not limited to Short Form (36) Health Survey and Barthel Index of Activities of Daily Living will not be performed, which will be considered in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with avascular necrosis of the femoral head diagnosed according to the previous criteria: Bone nonunion as indicated by a clear fracture line on X-ray images 12 months after femoral neck fracture; cystic degeneration, sclerosis, and uneven density on X-ray images and CT scans
* Patients with osteoporosis diagnosed according to a previous report: Bone density T value < -2.5 or bone mass decrease by 25%
* Patients with femoral neck fracture diagnosed according to the previous criteria (Chen and Wang, 2013): Presence of a fracture line on anterior- posterior X-ray images of the hip joint, and CT and MRI examination in combination with clinical symptoms and physical sign are necessary if no fracture line appears
* Age 60-80 years
* Healthy and able to tolerate anesthesia and surgery
* Provision of informed consent about participation and trial procedure

Exclusion Criteria:

* Alcohol abuse or long-term use of hormone drugs
* Infection of tissue around the hip joint
* Bone metabolism disorders other than osteoporosis, such as renal osteodystrophy and osteomalacia
* Heart, lung, brain, or other systemic diseases
* Advanced malignant tumor
* Recent cerebral hemorrhage, myocardial infarction, or failure of important organs
* Injured limb with deep venous thrombosis
* Inability to tolerate surgery

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes of Harris hip scores | at baseline, 1, 6 and 12 months after surgery
  To evaluate the recovery of hip joint function from the domains covering pain, function, absence of deformity, and range of motion, with higher scores indicating better hip joint function. Hip joint function is scored as follows: ≥ 90 is excellent, 80-89 very good, 70-79 good, and < 70 poor.

SECONDARY OUTCOMES:
Changes of VAS scores | at baseline, 1, 6 and 12 months after surgery
  To evaluate the severity of pain and ranges from 0-10, with higher scores indicating more severe pain. A score of 0 represents no pain, scores > 0 and ≤ 3 represent mild pain, scores > 3 and ≤ 6 moderate pain, and scores > 6 and ≤ 10 severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Ren, Master, Principal Investigator — Affiliated Hospital of Qinghai University

IPD SHARING:
Plan to Share IPD: Undecided